CLINICAL TRIAL: NCT01972789
Title: A Phase IV, Randomised, Single Masked Study Investigating the Efficacy and Safety of Ranibizumab "Inject and Extend" Using an Intensive Retinal Fluid Retreatment Regimen Compared to a Relaxed Retinal Fluid Retreatment Regimen in Patients With Wet Age-related Macular Degeneration (AMD)
Brief Title: Comparison of Treatment Regimens Using Ranibizumab: Intensive (Resolution of Intra- and Sub-retinal Fluid) vs Relaxed (Resolution of Intra-retinal Fluid and/or Sub-retinal Fluid >200µm at the Foveal Centre)
Acronym: FLUID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002AAU15
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-09

CONDITIONS: Subfoveal Choroidal Neovascularization CNV Secondary to Wet Age-related Macular Degeneration AMD
Keywords: Subfoveal choroidal neovascularization (CNV); wet age-related macular degeneration(AMD); inject and extend; retinal fluid
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive retinal fluid regimen (Experimental): Ranibizumab 0.5mg is given monthly for the first 3 months followed by an individualised treatment regimen as determined by disease activity defined by a loss of ≥5 letters, new retinal haemorrhage, presence of any IRF or SRF on OCT.
  Interventions: Drug: Ranibizumab
- Relaxed retinal fluid regimen (Experimental): Ranibizumab 0.5mg is given monthly for the first 3 months followed by an individualised treatment regimen as determined by disease activity defined by a loss of ≥5 letters, new retinal haemorrhage, presence of IRF or SRF >200 um on OCT.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab solution for injection is commercially supplied in two presentations: as a pre-filled syringe (containing 1.65 mg of ranibizumab in 0.165 mL solution) and as a vial (containing 2.3 mg of ranibizumab in 0.23 mL solution) corresponding to a recommended dose of 0.5 mg (0.05 mL) given as a single intravitreal injection. It will be prescribed and administered by the investigator or designee
  Other Names: LUCENTIS

SUMMARY:
To evaluate and compare two individualised ranibizumab treatment regimens, differentiated by the definition of disease activity, which determines the treatment interval until the next injection. The results will be used to generate recommendations about ranibizumab treatment when using an 'inject and extend' approach to maximise patient outcomes, while reducing the need for potentially unnecessary intravitreal injections. This study will also investigate if genotypic expression influences response to intravitreal injections of ranibizumab between the two treatment arms.

The study hypothesis is that intravitreal ranibizumab when administered to resolve IRF (and/or SRF >200 μm at the foveal centre) results in visual acuity benefit that is not clinically worse than intravitreal ranibizumab when administered to completely resolve both IRF and SRF in patients with wet AMD

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of subfoveal CNV secondary to wet AMD without restriction of lesion size, with visual impairment being exclusively due to an active wet AMD lesion. Active lesions will be characterised by any of the following: abnormal retinal thickness, with evidence of intraretinal, subretinal or sub-pigment epithelial fluid accumulation, confirmed by OCT; presence of intraretinal or subretinal haemorrhage; new leakage shown on a FA; CNV enlargement on FA unless solely due to dry, fibrotic staining; visual acuity deterioration considered likely to represent CNV.
2. BCVA score at both Screening and Baseline must be 23 letters or more as measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR charts (a Snellen visual acuity or equivalent of 20/320 or more may be used as an alternative at Screening).

Exclusion Criteria:

1. Any active periocular or ocular infection or inflammation (e.g., blepharitis, conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) at the time of Screening or Baseline.
2. Uncontrolled glaucoma (intraocular pressure [IOP] ≥30 mm Hg on medication) at the time of Screening or Baseline.
3. Neovascularisation of the iris or neovascular glaucoma at the time of Screening or Baseline.
4. Visually significant cataract, aphakia, severe vitreous haemorrhage, rhegmatogenous retinal detachment, proliferative diabetic retinopathy or CNV of any cause other than wet AMD at the time of screening and baseline.
5. Structural damage within 0.5 disc diameter of the centre of the macula (e.g., vitreomacular traction, epiretinal membrane, scar, laser burn, foveal atrophy) at the time of screening that in the investigator's opinion could preclude visual function improvement with treatment.
6. Treatment with any anti-angiogenic drugs (including any anti-VEGF agents) prior to Baseline in study eye (allowed in fellow eye).
7. Any intraocular procedure (including Ytrium-Aluminium- Garnet capsulotomy) within 2 months prior to Baseline or anticipated within the next 6 months following Baseline in th study eye (allowed in fellow eye).

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Australia (15):
  - Novartis Investigative Site, Albury, New South Wales
  - Novartis Investigative Site, Chatswood, New South Wales
  - Novartis Investigative Site, Eastwood, New South Wales
  - Novartis Investigative Site, Hurtsville, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, North Ryde, New South Wales
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Strathfield, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, South Launceston, Tasmania
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arnold JJ, Markey CM, Kurstjens NP, Guymer RH. The role of sub-retinal fluid in determining treatment outcomes in patients with neovascular age-related macular degeneration--a phase IV randomised clinical trial with ranibizumab: the FLUID study. BMC Ophthalmol. 2016 Mar 24;16:31. doi: 10.1186/s12886-016-0207-3. PMID 27009515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: a total of 349 subjects were randomized to the study (intensive arm, 174; relaxed arm, 175). relaxed 173).
Pre-assignment Details: Two randomized subjects, 1 in each treatment group, did not receive study treatment and were excluded from the safety set (347 subjects: intensive arm, 173; relaxed arm, 174). 2 subjects did not have correctly measured BCVA at baseline and were excluded from the FAS (345 subjects: intensive 172;
Period: Overall Study
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Started | 174 | 175
Completed | 134 | 145
Not Completed | 40 | 30
Not completed — Adverse Event | 11 | 4
Not completed — Subject withdrew consent | 14 | 12
Not completed — Lost to Follow-up | 4 | 7
Not completed — Death | 7 | 5
Not completed — Protocol deviation | 1 | 0
Not completed — Physician Decision | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen | Total
Number analyzed (Participants) | 174 | 175 | 349
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.3 (8.12) | 78.8 (8.17) | 79 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 89 | 189
  Male | 74 | 86 | 160
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 163 | 171 | 334
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best-corrected Visual Acuity (BCVA) From Baseline to 24 Months.
Description: Best-corrected visual acuity (BCVA) with refraction will be taken using a logMAR chart at a distance of 3 metres in the study eye at baseline and month 24.
Time Frame: Baseline to month 24
Population: Full Analysis Set (FAS): The Full Analysis Set (FAS) compromises all subjects randomised and whom have at least one post-Baseline efficacy value for the primary endpoint
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
Letters | 3.2 (16.51) | 2.5 (16.56)
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Test type: Non-Inferiority — This is a non-inferiority study design, with a pre-specified non-inferiority margin of 5 letters between intensive and relaxed groups. That is, if the change from Baseline in BCVA at Month 24 in the intensive group is not more than 5 letters higher than the relaxed group, then the relaxed group is regarded not inferior to the intensive group; p = 0.787, Mixed Models Analysis; Odds Ratio (OR) = 0.40, 95% CI 2-sided [-2.51 to 3.32]

2. Secondary Outcome: Mean Change in BCVA From Baseline to Month 12.
Description: Best-corrected visual acuity (BCVA) with refraction will be taken using a logMAR chart at a distance of 3 metres in the study eye at baseline and month 12.
Time Frame: Baseline to month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
Letters | 4.6 (14.69) | 3.9 (12.73)
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Test type: Other; p = 0.833, Mixed Models Analysis; Odds Ratio (OR) = -0.31, 95% CI 2-sided [-3.20 to 2.58]

3. Secondary Outcome: Mean Change in Central Retinal Thickness (CRT) From Baseline to Month 12 and 24.
Description: Central retinal thickness will be measured by Optical Coherence Tomography (OCT) at every visit.
Time Frame: Baseline to month 12 and month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
μm
  Month 12: number analyzed (Participants) | 154 | 150
  Month 12 | -147.1 (168.33) | -125.6 (133.08)
  Month 24: number analyzed (Participants) | 141 | 145
  Month 24 | -158.9 (170.44) | -126.9 (140.01)
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Test type: Other; p = 0.054, Mixed Models Analysis; Odds Ratio (OR) = -21.39, 95% CI 2-sided [-43.17 to 0.39]

4. Secondary Outcome: Mean Number of Injections From Baseline to Month 12 and 24
Description: The number of injections will be determined by the individual patient response to ranibizumab therapy and potential for extension between injections based on specific criteria: loss of visual acuity, new retinal haemorrhage, and presence of IRF or SRF on OCT.
Time Frame: Baseline to month 12 to month 24.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Injections
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
Injections
  Month 12 | 9.5 (2.60) | 8.9 (2.25)
  Month 24 | 17 (6.48) | 15.8 (5.91)
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Test type: Other; p = 0.001, Mixed Model; Negative Binomial Regression = 1.11, 95% CI 2-sided [1.04 to 1.18]

5. Secondary Outcome: Mean Change in Area of New and Existing Geographic Atrophy From Baseline to Month 12 and 24.
Description: Autofluorescence will be measured by multimodal imaging to assess the presence and development of geographic atrophy in the study at baseline, and month 12 and 24.
Time Frame: Baseline to months 12 and 24.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
mm^2
  Month 12: number analyzed (Participants) | 149 | 150
  Month 12 | 0.8 (2.13) | 0.7 (1.80)
  Month 24: number analyzed (Participants) | 132 | 139
  Month 24 | 1.5 (3.18) | 1.2 (2.62)
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Test type: Other; p = 0.338, Mixed Models Analysis; Odds Ratio (OR) = 0.26, 95% CI 2-sided [-0.28 to 0.80]

6. Secondary Outcome: Proportion of Patients Showing Newly Developed Geographic Atrophy (GA) at Months 12 and 24
Description: A multimodal imaging approach will be used to assess the presence of new geographic atrophy (defined as incorporating both geographic atrophy and atrophy associated with the CNV) in the study eye at baseline, and month 12 and 24. Image modalities will include fundus autofluorescence (AF) imaging, infrared imaging, OCT and colour fundus (CF) photographs. Atrophy will be diagnosed if FA and one other modality confirm the presence of macular atrophy
Time Frame: Months 12 and 24
Population: Full Analysis Set (FAS): The Full Analysis Set (FAS) compromises all subjects randomized and whom have at least one post-Baseline efficacy value for the primary endpoint
Measure: Number; unit: Participants
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
Participants
  Month 12, GA present: number analyzed (Participants) | 128 | 128
  Month 12, GA present | 25 | 18
  Month 12, GA absent: number analyzed (Participants) | 128 | 128
  Month 12, GA absent | 103 | 110
  Month 24, GA present: number analyzed (Participants) | 112 | 123
  Month 24, GA present | 32 | 29
  Month 24, GA absent: number analyzed (Participants) | 112 | 123
  Month 24, GA absent | 80 | 94
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Month 12; Test type: Other; p = 0.284, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.74 to 2.80]
Statistical Analysis 2: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Month 24; Test type: Other; p = 0.407, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.71 to 2.33]

7. Secondary Outcome: Proportion of Patients Showing no IRF and SRF at Months 2, 12 and 24.
Description: Assessed by Optical Coherence Tomography (OCT) and confirmed by a central reading centre.
Time Frame: Months 2, 12 and 24.
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
Participants
  Month 2: number analyzed (Participants) | 170 | 172
  Month 2 | 106 | 93
  month 12: number analyzed (Participants) | 154 | 152
  month 12 | 87 | 72
  Month 24: number analyzed (Participants) | 141 | 146
  Month 24 | 64 | 56
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Test type: Other; p = 0.217, Regression, Logistic; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.12 to 1.04]

8. Secondary Outcome: Proportion of Patients Showing Greater Than or Equal to 15 Letters Early Treatment Diabetic Retinopathy (ETDRS) Gain From Baseline to Month 12 and 24.
Description: Best-corrected visual acuity (BCVA) with refraction will be taken using a logMAR chart at a distance of 3 metres in the study eye at baseline and months 2, 12 and 24.
Time Frame: Baseline to months 12 and 24.
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
Participants
  Month 12: number analyzed (Participants) | 154 | 155
  Month 12 | 29 | 24
  Month 24: number analyzed (Participants) | 147 | 151
  Month 24 | 25 | 24
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Test type: Other; p = 0.615, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.42 to 1.66]

9. Secondary Outcome: Proportion of Patients Showing Less Than 15 Letters ETDRS Loss From Baseline to Month 12 and 24.
Description: Best-corrected visual acuity with refraction will be taken using a logMAR chart at a distance of 3 metres in the study eye at baseline and months 2, 12 and 24.
Time Frame: Baseline to months 12 and 24
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
Participants
  Month 12: number analyzed (Participants) | 154 | 155
  Month 12 | 142 | 141
  Month 24: number analyzed (Participants) | 147 | 151
  Month 24 | 129 | 132
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Test type: Other; p = 0.819, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.54 to 2.18]

10. Secondary Outcome: Number of Participants With the Genotypes Associated With Age-Related Macular Degeneration (AMD) and Response to Treatment at Baseline; Correlation With Visual Acuity (VA) Outcome and Ability to Dry the Retina.
Description: DNA will be extracted from saliva and genotyping performed on the significantly associated single nucleotide polymorphisms (SNPs) identified by the AMD Gene Consortium (Nature Genetics, March 2013). Genotypes will be derived through the use of a Sequenom Iplex protocol. No correlation analyses were performed.
Time Frame: Baseline or following consent
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
Participants
  RS10490924 GG: number analyzed (Participants) | 124 | 127
  RS10490924 GG | 44 | 47
  RS10490924 GT: number analyzed (Participants) | 124 | 127
  RS10490924 GT | 56 | 57
  RS10490924 TT: number analyzed (Participants) | 124 | 127
  RS10490924 TT | 24 | 23
  RS1061170 CC: number analyzed (Participants) | 125 | 125
  RS1061170 CC | 35 | 43
  RS1061170 CT: number analyzed (Participants) | 125 | 125
  RS1061170 CT | 61 | 61
  RS1061170 TT: number analyzed (Participants) | 125 | 125
  RS1061170 TT | 29 | 21
  RS10737680 AA: number analyzed (Participants) | 125 | 127
  RS10737680 AA | 68 | 82
  RS10737680 AC: number analyzed (Participants) | 125 | 127
  RS10737680 AC | 48 | 37
  RS10737680 CC: number analyzed (Participants) | 125 | 127
  RS10737680 CC | 9 | 8
  RS11200638 AA: number analyzed (Participants) | 125 | 127
  RS11200638 AA | 21 | 23
  RS11200638 AG: number analyzed (Participants) | 125 | 127
  RS11200638 AG | 58 | 58
  RS11200638 GG: number analyzed (Participants) | 125 | 127
  RS11200638 GG | 46 | 46
  RS121913059 CC: number analyzed (Participants) | 125 | 127
  RS121913059 CC | 124 | 127
  RS121913059 CT: number analyzed (Participants) | 125 | 127
  RS121913059 CT | 1 | 0
  RS13278062 GG: number analyzed (Participants) | 125 | 127
  RS13278062 GG | 29 | 17
  RS13278062 GT: number analyzed (Participants) | 125 | 127
  RS13278062 GT | 60 | 75
  RS13278062 TT: number analyzed (Participants) | 125 | 127
  RS13278062 TT | 36 | 35
  RS141853578 CC: number analyzed (Participants) | 125 | 127
  RS141853578 CC | 125 | 125
  RS147859257 GT: number analyzed (Participants) | 125 | 127
  RS147859257 GT | 2 | 1
  RS147859257 TT: number analyzed (Participants) | 125 | 127
  RS147859257 TT | 123 | 126
  RS1864163 AA: number analyzed (Participants) | 123 | 126
  RS1864163 AA | 9 | 7
  RS1864163 AG: number analyzed (Participants) | 123 | 126
  RS1864163 AG | 29 | 46
  RS1864163 GG: number analyzed (Participants) | 123 | 126
  RS1864163 GG | 85 | 73
  RS2230199 CC: number analyzed (Participants) | 124 | 127
  RS2230199 CC | 81 | 67
  RS2230199 CG: number analyzed (Participants) | 124 | 127
  RS2230199 CG | 37 | 52
  RS2230199 GG: number analyzed (Participants) | 124 | 127
  RS2230199 GG | 6 | 8
  RS3130783 AA: number analyzed (Participants) | 125 | 127
  RS3130783 AA | 77 | 91
  RS3130783 AG: number analyzed (Participants) | 125 | 127
  RS3130783 AG | 44 | 32
  RS3130783 GG: number analyzed (Participants) | 125 | 127
  RS3130783 GG | 4 | 4
  RS334353 GG: number analyzed (Participants) | 125 | 127
  RS334353 GG | 6 | 11
  RS334353 GT: number analyzed (Participants) | 125 | 127
  RS334353 GT | 41 | 45
  RS334353 TT: number analyzed (Participants) | 125 | 127
  RS334353 TT | 78 | 71
  RS3812111 AA: number analyzed (Participants) | 124 | 122
  RS3812111 AA | 31 | 16
  RS3812111 AT: number analyzed (Participants) | 124 | 122
  RS3812111 AT | 57 | 52
  RS3812111 TT: number analyzed (Participants) | 124 | 122
  RS3812111 TT | 36 | 54
  RS429608 AA: number analyzed (Participants) | 124 | 123
  RS429608 AA | 2 | 1
  RS429608 AG: number analyzed (Participants) | 124 | 123
  RS429608 AG | 19 | 19
  RS429608 GG: number analyzed (Participants) | 124 | 123
  RS429608 GG | 103 | 103
  RS4420638 AA: number analyzed (Participants) | 124 | 127
  RS4420638 AA | 89 | 96
  RS4420638 AG: number analyzed (Participants) | 124 | 127
  RS4420638 AG | 35 | 31
  RS4698775 GG: number analyzed (Participants) | 124 | 126
  RS4698775 GG | 11 | 8
  RS4698775 GT: number analyzed (Participants) | 124 | 126
  RS4698775 GT | 53 | 71
  RS4698775 TT: number analyzed (Participants) | 124 | 126
  RS4698775 TT | 60 | 47
  RS5749482 CC: number analyzed (Participants) | 125 | 127
  RS5749482 CC | 4 | 1
  RS5749482 CG: number analyzed (Participants) | 125 | 127
  RS5749482 CG | 26 | 26
  RS5749482 GG: number analyzed (Participants) | 125 | 127
  RS5749482 GG | 95 | 100
  RS6795735 CC: number analyzed (Participants) | 124 | 127
  RS6795735 CC | 43 | 37
  RS6795735 CT: number analyzed (Participants) | 124 | 127
  RS6795735 CT | 53 | 63
  RS6795735 TT: number analyzed (Participants) | 124 | 127
  RS6795735 TT | 28 | 27
  RS8017304 AA: number analyzed (Participants) | 125 | 127
  RS8017304 AA | 57 | 65
  RS8017304 AG: number analyzed (Participants) | 125 | 127
  RS8017304 AG | 53 | 51
  RS8017304 GG: number analyzed (Participants) | 125 | 127
  RS8017304 GG | 15 | 11
  RS8135665 CC: number analyzed (Participants) | 124 | 127
  RS8135665 CC | 68 | 79
  RS8135665 CT: number analyzed (Participants) | 124 | 127
  RS8135665 CT | 50 | 41
  RS8135665 TT: number analyzed (Participants) | 124 | 127
  RS8135665 TT | 6 | 7
  RS920915 CC: number analyzed (Participants) | 124 | 127
  RS920915 CC | 32 | 33
  RS920915 CG: number analyzed (Participants) | 124 | 127
  RS920915 CG | 64 | 60
  RS920915 GG: number analyzed (Participants) | 124 | 127
  RS920915 GG | 28 | 34
  RS943080 CC: number analyzed (Participants) | 124 | 127
  RS943080 CC | 27 | 35
  RS943080 CT: number analyzed (Participants) | 124 | 127
  RS943080 CT | 57 | 64
  RS943080 TT: number analyzed (Participants) | 124 | 127
  RS943080 TT | 40 | 28
  RS9542236 CC: number analyzed (Participants) | 125 | 127
  RS9542236 CC | 26 | 26
  RS9542236 CT: number analyzed (Participants) | 125 | 127
  RS9542236 CT | 61 | 63
  RS9542236 TT: number analyzed (Participants) | 125 | 127
  RS9542236 TT | 38 | 38

11. Secondary Outcome: Proportion of Patients With Both SRF (Sub-retinal Fluid) and IRF (Intra-retinal Fluid) Who Despite Monthly Treatment do Not Resolve Their SRF
Description: Assessed by Optical Coherence Tomography (OCT) and confirmed by a central reading centre.
Time Frame: Month 12 and 24
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 6 | 6
Participants
  Month 12: number analyzed (Participants) | 6 | 3
  Month 12 | 3 | 2
  Month 24: number analyzed (Participants) | 2 | 4
  Month 24 | 1 | 2
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Test type: Other; p = 0.565, Regression, Logistic; Odds Ratio (OR) = 4.32, 95% CI 2-sided [0.03 to 630.5]

12. Secondary Outcome: The Number of Times a Participant Needs to Return to Monthly Treatments During the 24 Months.
Description: Treatment requirements will be determined by the individual patient disease activity as measured by OCT, BCVA, colour fundus photography and fluorescein angiography (FA). Analysis was not performed.
Time Frame: Month 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Intensive Retinal Fluid Regimen | Relaxed Retinal Fluid Regimen
Number analyzed (Participants) | 172 | 173
Visits | 10.6 (8.34) | 7.6 (8.09)
Statistical Analysis 1: Comparison: Intensive Retinal Fluid Regimen vs Relaxed Retinal Fluid Regimen; Test type: Other; p = 0.034, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.03 to 1.90]

ADVERSE EVENTS:
Time Frame: Up to 24 month
Description: AE additional description
Groups:
- Intensive: Intensive
- Relaxed: Relaxed
Arm/Group | Intensive | Relaxed
All-Cause Mortality (participants affected / at risk) | 7/173 | 5/174
Serious Adverse Events (participants affected / at risk) | 58/173 | 58/174
Other Adverse Events (participants affected / at risk) | 109/173 | 114/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive (N=173) | Relaxed (N=174)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 7
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Macular hole (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Retinal pigment epithelial tear (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal oedema (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Catheter site extravasation (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 2 | 2
Disease progression (General disorders) | 1 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 2 | 0
Endophthalmitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Klebsiella infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 3
Pertussis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 10 | 5
Sepsis (Infections and infestations) | 0 | 1
Skin graft infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Blood sodium decreased (Investigations) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 4
Convulsion (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 4 | 2
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 1 | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 1 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 2
Anaemia(Non-ocular) (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia(Non-ocular) (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia(Non-ocular) (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction(Non-ocular) (Cardiac disorders) | 1 | 2
Arrhythmia(Non-ocular) (Cardiac disorders) | 0 | 1
Atrial fibrillation(Non-ocular) (Cardiac disorders) | 2 | 7
Bradycardia(Non-ocular) (Cardiac disorders) | 0 | 1
Cardiac failure congestive(Non-ocular) (Cardiac disorders) | 1 | 0
Cardiac failure(Non-ocular) (Cardiac disorders) | 2 | 1
Cardiogenic shock(Non-ocular) (Cardiac disorders) | 0 | 1
Coronary artery disease(Non-ocular) (Cardiac disorders) | 0 | 1
Myocardial infarction(Non-ocular) (Cardiac disorders) | 1 | 1
Myocardial ischaemia(Non-ocular) (Cardiac disorders) | 1 | 0
Pericarditis(Non-ocular) (Cardiac disorders) | 0 | 1
Tachycardia(Non-ocular) (Cardiac disorders) | 0 | 1
Ventricular tachycardia(Non-ocular) (Cardiac disorders) | 1 | 0
Phimosis(Non-ocular) (Congenital, familial and genetic disorders) | 0 | 1
Meniere's disease(Non-ocular) (Ear and labyrinth disorders) | 1 | 0
Vertigo positional(Non-ocular) (Ear and labyrinth disorders) | 0 | 1
Macular hole(Left eye) (Eye disorders) | 0 | 1
Retinal artery occlusion(Right eye) (Eye disorders) | 1 | 0
Retinal pigment epithelial tear(Left eye) (Eye disorders) | 0 | 1
Abdominal pain upper(Non-ocular) (Gastrointestinal disorders) | 0 | 1
Alcoholic pancreatitis(Non-ocular) (Gastrointestinal disorders) | 0 | 1
Barrett's oesophagus(Non-ocular) (Gastrointestinal disorders) | 1 | 0
Dysphagia(Non-ocular) (Gastrointestinal disorders) | 1 | 0
Gastric ulcer(Non-ocular) (Gastrointestinal disorders) | 1 | 0
Gastrointestinal oedema(Non-ocular) (Gastrointestinal disorders) | 1 | 0
Haematemesis(Non-ocular) (Gastrointestinal disorders) | 0 | 1
Intestinal perforation(Non-ocular) (Gastrointestinal disorders) | 1 | 0
Pancreatitis(Non-ocular) (Gastrointestinal disorders) | 0 | 1
Peptic ulcer(Non-ocular) (Gastrointestinal disorders) | 0 | 1
Vomiting(Non-ocular) (Gastrointestinal disorders) | 1 | 0
Catheter site extravasation(Non-ocular) (General disorders) | 0 | 1
Chest pain(Non-ocular) (General disorders) | 1 | 1
Death(Non-ocular) (General disorders) | 2 | 2
Disease progression(Non-ocular) (General disorders) | 1 | 2
Cholecystitis acute(Non-ocular) (Hepatobiliary disorders) | 0 | 2
Cholecystitis chronic(Non-ocular) (Hepatobiliary disorders) | 0 | 1
Cholelithiasis(Non-ocular) (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis(Non-ocular) (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic(Non-ocular) (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity(Non-ocular) (Immune system disorders) | 0 | 1
Appendicitis(Non-ocular) (Infections and infestations) | 0 | 1
Arthritis infective(Non-ocular) (Infections and infestations) | 1 | 0
Bacteraemia(Non-ocular) (Infections and infestations) | 0 | 1
Bronchitis(Non-ocular) (Infections and infestations) | 1 | 0
Cystitis() (Infections and infestations) | 1 | 0
Cystitis(Non-ocular) (Infections and infestations) | 1 | 0
Endophthalmitis(Right eye) (Infections and infestations) | 1 | 0
Escherichia bacteraemia(Non-ocular) (Infections and infestations) | 0 | 1
Gastroenteritis viral(Non-ocular) (Infections and infestations) | 1 | 0
Gastroenteritis(Non-ocular) (Infections and infestations) | 1 | 1
Herpes zoster(Non-ocular) (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease(Non-ocular) (Infections and infestations) | 1 | 0
Influenza(Non-ocular) (Infections and infestations) | 2 | 0
Klebsiella infection(Non-ocular) (Infections and infestations) | 0 | 1
Localised infection(Non-ocular) (Infections and infestations) | 0 | 1
Lower respiratory tract infection(Non-ocular) (Infections and infestations) | 1 | 3
Pertussis(Left eye) (Infections and infestations) | 1 | 0
Pneumonia(Non-ocular) (Infections and infestations) | 10 | 5
Sepsis(Non-ocular) (Infections and infestations) | 0 | 1
Skin graft infection(Non-ocular) (Infections and infestations) | 1 | 0
Urinary tract infection(Non-ocular) (Infections and infestations) | 1 | 2
Urosepsis(Non-ocular) (Infections and infestations) | 0 | 1
Accidental overdose(Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Cataract operation complication(Right eye) (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture(Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Fall(Non-ocular) (Injury, poisoning and procedural complications) | 4 | 2
Femoral neck fracture(Non-ocular) (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture(Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Head injury(Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture(Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture(Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation(Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Joint injury(Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Laceration(Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture(Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary contusion(Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture(Non-ocular) (Injury, poisoning and procedural complications) | 2 | 0
Skull fracture(Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm(Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Blood sodium decreased(Non-ocular) (Investigations) | 1 | 0
Fluid overload(Non-ocular) (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia(Non-ocular) (Metabolism and nutrition disorders) | 2 | 0
Back pain(Non-ocular) (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia(Non-ocular) (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome(Non-ocular) (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ductal adenocarcinoma of pancreas(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal carcinoma(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lung neoplasm malignant(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to abdominal cavity(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of lung(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma(Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cerebral haemorrhage(Non-ocular) (Nervous system disorders) | 1 | 0
Cerebrovascular accident(Non-ocular) (Nervous system disorders) | 3 | 4
Convulsion(Non-ocular) (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type(Non-ocular) (Nervous system disorders) | 1 | 0
Dizziness(Non-ocular) (Nervous system disorders) | 0 | 1
Neuralgia(Non-ocular) (Nervous system disorders) | 0 | 1
Presyncope(Non-ocular) (Nervous system disorders) | 1 | 0
Syncope(Non-ocular) (Nervous system disorders) | 2 | 0
Transient ischaemic attack(Non-ocular) (Nervous system disorders) | 4 | 2
Confusional state(Non-ocular) (Psychiatric disorders) | 1 | 0
Delirium(Non-ocular) (Psychiatric disorders) | 1 | 0
Haematuria(Non-ocular) (Renal and urinary disorders) | 1 | 1
Nephrolithiasis(Non-ocular) (Renal and urinary disorders) | 1 | 0
Renal disorder(Non-ocular) (Renal and urinary disorders) | 1 | 0
Renal failure acute(Non-ocular) (Renal and urinary disorders) | 0 | 1
Renal impairment(Non-ocular) (Renal and urinary disorders) | 1 | 0
Renal injury(Non-ocular) (Renal and urinary disorders) | 0 | 1
Urinary retention(Non-ocular) (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema(Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma(Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease(Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax(Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism(Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis(Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension(Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer(Non-ocular) (Skin and subcutaneous tissue disorders) | 0 | 1
Hospitalisation() (Surgical and medical procedures) | 0 | 1
Hospitalisation(Non-ocular) (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention(Non-ocular) (Surgical and medical procedures) | 0 | 1
Arteriovenous fistula(Non-ocular) (Vascular disorders) | 1 | 0
Blood pressure fluctuation(Non-ocular) (Vascular disorders) | 0 | 1
Haemorrhage(Non-ocular) (Vascular disorders) | 0 | 1
Hypertension(Non-ocular) (Vascular disorders) | 0 | 1
Hypotension(Non-ocular) (Vascular disorders) | 1 | 0
Orthostatic hypotension(Non-ocular) (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive (N=173) | Relaxed (N=174)
Age-related macular degeneration (Eye disorders) | 18 | 17
Cataract (Eye disorders) | 4 | 13
Conjunctival haemorrhage (Eye disorders) | 8 | 13
Dry eye (Eye disorders) | 8 | 9
Eye pain (Eye disorders) | 28 | 24
Eye pruritus (Eye disorders) | 9 | 5
Foreign body sensation in eyes (Eye disorders) | 8 | 11
Lacrimation increased (Eye disorders) | 17 | 8
Retinal haemorrhage (Eye disorders) | 7 | 12
Vision blurred (Eye disorders) | 16 | 10
Visual acuity reduced (Eye disorders) | 9 | 11
Vitreous detachment (Eye disorders) | 11 | 11
Vitreous floaters (Eye disorders) | 21 | 11
Nausea (Gastrointestinal disorders) | 8 | 10
Disease progression (General disorders) | 9 | 6
Injection site pain (General disorders) | 14 | 8
Influenza (Infections and infestations) | 26 | 16
Lower respiratory tract infection (Infections and infestations) | 10 | 11
Nasopharyngitis (Infections and infestations) | 23 | 29
Urinary tract infection (Infections and infestations) | 11 | 13
Fall (Injury, poisoning and procedural complications) | 21 | 15
Dizziness (Nervous system disorders) | 11 | 9
Headache (Nervous system disorders) | 16 | 9
Depression (Psychiatric disorders) | 3 | 11
Cataract operation (Surgical and medical procedures) | 6 | 10
Age-related macular degeneration(Left eye) (Eye disorders) | 8 | 14
Age-related macular degeneration(Right eye) (Eye disorders) | 11 | 5
Cataract(Left eye) (Eye disorders) | 2 | 9
Eye pain(Left eye) (Eye disorders) | 12 | 11
Eye pain(Right eye) (Eye disorders) | 11 | 13
Lacrimation increased(Right eye) (Eye disorders) | 9 | 4
Retinal haemorrhage(Left eye) (Eye disorders) | 6 | 9
Vision blurred(Right eye) (Eye disorders) | 9 | 3
Vitreous floaters(Left eye) (Eye disorders) | 14 | 5
Nausea(Non-ocular) (Gastrointestinal disorders) | 8 | 10
Injection site pain(Right eye) (General disorders) | 9 | 4
Influenza(Non-ocular) (Infections and infestations) | 26 | 16
Lower respiratory tract infection(Non-ocular) (Infections and infestations) | 10 | 11
Nasopharyngitis(Non-ocular) (Infections and infestations) | 23 | 29
Urinary tract infection(Non-ocular) (Infections and infestations) | 11 | 13
Fall(Non-ocular) (Injury, poisoning and procedural complications) | 21 | 15
Dizziness(Non-ocular) (Nervous system disorders) | 11 | 9
Headache(Non-ocular) (Nervous system disorders) | 15 | 8
Depression(Non-ocular) (Psychiatric disorders) | 3 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT01972789/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT01972789/SAP_001.pdf